CLINICAL TRIAL: NCT06487650
Title: The Development and Evaluation of Sleep Intervention for Perinatal Family
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: N202204079
Record Dates: First submitted 2024-06-13; First posted 2024-07-05 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Sleep; Psychological Distress; Perinatal Problems
Keywords: sleep quality; perinatal; depression; anxiety; infant sleep; infant health
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleep intervention (Experimental): Participants in the intervention group will receive both the standardized usual care and the sleep intervention. The intervention consists of sleep education, health professional support, and counseling. The intervention will be delivered from pregnancy to postpartum for mothers and fathers.
  Interventions: Behavioral: sleep intervention
- Control (Active Comparator): Participants in the control group will receive a perinatal health booklet in addition to the standardized usual care.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: sleep intervention — At the beginning of the intervention, participants will have an orientation and overview of the program. Then, participants will follow the curriculum of modules, and professional feedback to complete the intervention.
  Arms: sleep intervention
Behavioral: Control group — Participants in control group will follow standardized usual care and a perinatal health booklet
  Arms: Control

SUMMARY:
Background: Sleep disruptions and disturbances are highly prevalent among new mothers and fathers and negatively affect their mental health and infant development outcomes. Effective sleep interventions are vital for family health.

Objectives: To develop a sleep intervention for mother-father-infant triads, and to evaluate the effects on sleep improvement, emotional distress, and infant health outcomes.

Methods: In this proposal, we plan to conduct a parallel-group two-arm randomized controlled trial on pregnant women and their partners. Mother-father-infant triads will be recruited and randomly allocated to the intervention group (receiving a sleep intervention) or the control group. Data will be collected with repeated measures, and the relationship between studied variables will be analyzed with descriptive and inferential statistics.

Anticipatory results: The development and evaluation of an evidence-based sleep intervention will provide a scientific insight into sleep care for pregnant women and their families.

DETAILED DESCRIPTION:
The primary outcome is the severity of insomnia symptoms. The secondary outcomes of parents' sleep quality, objective sleep indicators, symptoms of depression and anxiety, and heart rate variability will be collected. Infant sleep quality, infant feeding, and infant health outcomes will also be assessed. Data will be analyzed using descriptive and inferential statistics.

ELIGIBILITY:
Inclusion Criteria:

1. First-time mothers and their partners aged 20 and older;
2. Currently 30 weeks gestation or more, singleton;
3. insomnia severity index score greater than 10;
4. living with a husband or partner;
5. Both women and their partners are willing to participate in and adhere to the research protocol;
6. be able to read and speak the Mandarin language

Exclusion Criteria:

1. sleep disorders, depression or anxiety disorders;
2. medical diseases with abnormal heart rate variability, or arrhythmia;
3. taking medicines that may affect the autonomic nervous system or
4. night shift workers;
5. obstetric complications, including gestational hypertension, preterm labor, labor complications, or postpartum complications;
6. infants with fetal deformity, or neonatal complications;
7. no access to Internet resources

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | baseline, at 36-weeks' gestation, 2-week postpartum, 1-month, 3-month,6-month, and 12-month postpartum
  The Chinese version of the Insomnia Severity Index (ISI) is used to measure the severity of insomnia symptoms, a higher score indicates more severe insomnia symptoms.

SECONDARY OUTCOMES:
Sleep quality | baseline, at 36-weeks' gestation, postpartum 1 month, 3 months, 6 months, and 12-months
  The 19-item Chinese version of the Pittsburgh Sleep Quality Index (PSQI), will be used to measure sleep quality and sleep disturbance, higher score indicates worse sleep quality
Sleep duration using actigraphy | baseline, postpartum 1 month, 3 months, and 6 months.
  The Actiwatch will be used to collect objective data of sleep duration
Sleep sleep onset latency using actigraphy | baseline, postpartum 1 month, 3 months, and 6 months.
  The Actiwatch will be used to collect objective data of sleep onset latency
Sleep efficacy using actigraphy | baseline, postpartum 1 month, 3 months, and 6 months.
  The Actiwatch will be used to collect objective data of sleep efficacy
Wake after sleep onset using actigraphy | baseline, postpartum 1 month, 3 months, and 6 months.
  The Actiwatch will be used to collect objective data of wake after sleep onset
Infants sleep Questionnaire | postpartum 1 month, 3 months, 6 months, and 12-months
  Parents will be asked to rate their infant's sleep quality using the 19-item Brief Infant Sleep Questionnaire-Revised (BISQ-R). The BISQ will be used to assess sleep duration, duration of sleep by circadian rhythm, and night-time awakenings
Depressive symptoms | baseline, at 36-weeks' gestation, postpartum 1 month, 3 months, 6 months, and 12-months
  Maternal and paternal depressive symptoms will be assessed using the Taiwanese version of the 10-item Edinburgh Postnatal Depression Scale (EPDS), a higher score indicated more severe symptoms.
Anxiety symptoms | baseline, at 36-weeks' gestation, postpartum 1 month, 3 months, 6 months, and 12-months
  The 20-item State Anxiety subscale of the State-Trait Anxiety Inventory (STAI) will be used to measure levels of anxiety symptoms in mothers and fathers, higher score presents more severe symptoms.
Heart rate variability (HRV) measures | at baseline, postpartum 1 month, 3 months, and 6 months
  The resting interbeat interval will be recorded
Infant weight | postpartum 3 months, 6 months, and 12-months
  Infants' body weight in gram will be measured by trained data collectors using an electronic scale specifically for infants
Infant height | postpartum 3 months, 6 months, and 12-months
  Infants' height in cm will be measured by trained data collectors using an electronic scale specifically for infants
Infant development | postpartum 3 months, 6 months, and 12-months
  Infant's social and emotional development will be assessed using the Taiwanese version of the Ages & Stages Questionnaires: Social-Emotional-2 (ASQ: SE-2).
Infant feeding | postpartum 1 month, 3 months, and 6 months, and 12 months
  Infant feeding methods will be measured using a self-report questionnaire. The feeding methods, including initiated breastfeeding within 24 hours after birth, and type of breastfeeding.
Satisfaction of sleep intervention | immediately after interventions
  A structured questionnaire with a 5-point Likert scale will be used to collect the level of satisfaction of the sleep intervention upon completion of programs.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Kuo, Phd, Principal Investigator — Taipei Medical University

IPD SHARING:
Plan to Share IPD: No